CLINICAL TRIAL: NCT01643707
Title: Registry to Improve the Adoption of Consensus Treatment Guidelines (IMPROVE Brady)
Acronym: IMPROVE Brady
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: IMPROVE Brady
Record Dates: First submitted 2012-06-28; First posted 2012-07-18 (Estimated); Results first posted 2021-09-17 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Sinus Node Dysfunction
Keywords: Sick Sinus Syndrome; Bradycardia
MeSH Terms: conditions — Sick Sinus Syndrome; Bradycardia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Phase I: Control
- Phase II: Treatment
  Interventions: Behavioral: Evidence based guidelines and tools

INTERVENTIONS:
Behavioral: Evidence based guidelines and tools — Education, guidelines, tools
  Groups: Phase II

SUMMARY:
Registry to Improve the Adoption of Consensus Treatment Guidelines (IMPROVE Brady)

DETAILED DESCRIPTION:
The study is expected to provide evidence to support claim(s) that:

* Education and process improvement initiatives can improve the diagnosis of and appropriate therapy application for sinus node dysfunction (SND)
* The quality improvement methods studied have general applicability and can be used by all centers
* Appropriate treatment minimizes caregiver burden
* Appropriate treatment improves quality of life (QOL) and functional status compared to pre-implant

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 18 years of age
* Patient's heart rate meets at least one of the following:

  * Patient has a sinus rate ≤ 50 OR a junctional escape rhythm no faster than 50
  * Patient has a history of exercise intolerance
* Patient complains of general fatigue, shortness of breath, shortness of breath with exertion, syncope, light headed dizziness, palpitations, lethargy, dyspnea OR malaise within the last 30 days that are not related to other discovered causes (such as untreated hypothyroidism or anemia).
* Patient (or patient's legally authorized representative) is willing and able to sign and date written Patient Consent Form/Patient Data Release Consent

Exclusion Criteria:

* Patient has type II 2nd degree AV block, High degree AV block (2:1, 3:1, 4:1 etc.) or 3rd degree AV block
* Patient has recent history of blood loss
* Patient has a medical history leading to suspicion of neurological disorder
* Patient has a history of Chronic Atrial Fibrillation
* Patient is enrolled or planning to participate in a concurrent drug and/or device study at any time during the course of this clinical study without documented pre-approval from the Medtronic study manager
* Patient is not expected to survive for 12 months
* Patient is anticipated to be unwilling or unable to comply with the clinical investigation plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with possible sinus node dysfunction
Sampling Method: Non-Probability Sample
Enrollment: 1342 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- Hospital General de Agudos, Buenos Aires, Argentina
- Bangladesh (2):
  - National Heart Foundation Hospital and Research Institute, Dhaka
  - United Hospital Limited, Dhaka
- India (8):
  - CARE Hospitals, Hyderabad, Andhra Pradesh
  - Care Insitute of Medical Sciences, Ahmedabad, Gujarat
  - RajaRajeswari Medical College & Hospital, Bangalore, Karnataka
  - Max Balaji Hospital, New Delhi, National Capital Territory of Delhi
  - Madras Medical Mission Institute of Cardiovascular Diseases, Chennai, Tamil Nadu
  - King George's Medical University, Lucknow, Uttar Pradesh
  - The Mission Hospital, Durgapur, West Bengal
  - Max Devki Devi Heart and Vascular Institute, Delhi
- Mexico (3):
  - Centro Medico Nacional de Occidente IMSS, Mexico City
  - Hospital Central Militar, Mexico City
  - UMAE Hospital de Cardiologia Centro Medico nacional Siglo XXI IMSS, Mexico City
- Peru (2):
  - Hospital Nacional Carlos Alberto Seguín Escobedo, Arequipa
  - Instituto Nacional Cardiovascular, Lima
- Russia (4):
  - Amur State Medical Academy, Amur, Amur Oblast
  - Chelyabinsk Federal Center of Cardiovascular Surgery, Chelyabinsk
  - Federal Center of Cardio-Vascular Surgery, Krasnoyarsk
  - Center of Modern Cardiology, Krasnoyarsk
- Casa de Galicia, Montevideo, Uruguay

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Phase I served as a control period during which physicians assessed and treated subjects per their site's standard care practice. In Phase 2, investigators completed an educational workshop, were given access to the IMPROVE Brady toolkit and encouraged to adapt tools from this kit to create a practice-specific process improvement implementation.
Groups:
- Phase I: Phase I served as a control period during which physicians assessed and treated subjects per their site's standard care practice.
- Phase II: In Phase 2, investigators completed an educational workshop, were given access to the IMPROVE Brady toolkit and encouraged to adapt tools from this kit to create a practice-specific process improvement implementation.
Period: Overall Study
Arm/Group | Phase I | Phase II
Started | 858 | 484
Completed | 823 | 470
Not Completed | 35 | 14

BASELINE CHARACTERISTICS:
Population: Phase 1, the control phase, we expect to obtain baseline measurements for key variables including the rate of SND diagnosis and the rate of implantation of an IPG in subjects with an SND diagnosis.2nd phase, the experimental phase, patients will have scheduled follow-up to collect questionnaire data if they are implanted with an IPG.
Groups:
- Phase I: Phase I served as a control period during which physicians assessed and treated subjects per their site's standard care practice. Phase I of the study was to understand the current pathways at hospital for SND patient screening & management.
- Phase II: In Phase II, investigators completed an educational workshop, were given access to the IMPROVE Brady toolkit and encouraged to adapt tools from this kit to create a practice-specific process improvement implementation. The toolkit included: a physician training seminar, a diagnostic algorithm, patient education materials, a list of available therapy options, and/or information regarding the benefits and risks associated with the therapy options.
- Total: Total of all reporting groups
Arm/Group | Phase I | Phase II | Total
Number analyzed (Participants) | 823 | 470 | 1293
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (16.0) | 57.9 (14.9) | 59.3 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 277 | 128 | 405
  Male | 546 | 342 | 888
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnic Origin: Subject/Physician Chose not to provide information | 2 | 0 | 2
  Race/Ethnic Origin: Not reportable per local laws or regulations | 1 | 0 | 1
  Race/Ethnic Origin: American Indian or Alaska Native | 0 | 0 | 0
  Race/Ethnic Origin: Asian | 59 | 106 | 165
  Race/Ethnic Origin: Black or African American | 0 | 0 | 0
  Race/Ethnic Origin: Hispanic or Latino | 163 | 0 | 163
  Race/Ethnic Origin: Native Hawaiian or Pacific Islander | 0 | 0 | 0
  Race/Ethnic Origin: White or Caucasian | 142 | 0 | 142
  Race/Ethnic Origin: Indian | 444 | 345 | 789
  Race/Ethnic Origin: Two or More Races | 1 | 0 | 1
  Race/Ethnic Origin: Other | 10 | 19 | 29
  Race/Ethnic Origin: Unknown/Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: The Absolute Change in the Proportion of Subjects Diagnosed With SND Before and After Intervention
Description: The absolute change in the proportion of subjects diagnosed with SND before and after intervention
Time Frame: Up to 1 year post enrollment
Population: Only sites in South Asia participated in both Phase 1 and Phase 2, as such those subjects were included for objective analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Control subjects in the South Asia Region.
- Phase 2: Treatment subjects in the South Asia Region
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 508 | 470
Participants | 368 | 409
Statistical Analysis 1: Comparison: Phase 1 vs Phase 2; Test type: Superiority — A chi-square test was performed to determine a difference between Phase 1 and Phase 2; p < 0.00001, Chi-squared

2. Primary Outcome: The Absolute Change in the Proportion of Subjects Receiving Indicated Therapy Before and After Intervention
Description: Outcome measure applies to subjects that receive a SND diagnosis
Time Frame: Up to 6 months post diagnosis
Population: Subjects with an SND diagnosis
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Control subjects in South Asia Region with an SND Diagnosis
- Phase 2: Treatment subjects in South Asia Region with an SND Diagnosis
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 368 | 409
Participants | 63 | 130
Statistical Analysis 1: Comparison: Phase 1 vs Phase 2; Test type: Equivalence — Chi-Square test used to show any difference between Phase 1 and Phase 2; p < 0.0001, Chi-squared

3. Secondary Outcome: The Proportion of Phase I Subjects Diagnosed With SND and the Number of Diagnoses That Result in Indicated Therapy
Description: Enrolled subjects only with an SND diagnosis were reassessed at 6 and 12 months post enrollment were reassessed for IPG therapy.
Time Frame: SND diagnosis assessed at 6 and 12 months of follow-up from enrollment until resulting IPG therapy
Population: Only subjects diagnosed in each phase with SND.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 368 | 409
Participants
  Subjects Diagnosed | 368 | 409
  Subjects Implanted | 63 | 130
Statistical Analysis 1: Comparison: Phase 1 vs Phase 2; Test type: Equivalence — Chi-Square test used to show any difference between Phase 1 and Phase 2; p < 0.0001, Chi-squared — This endpoint was covered in primary objective 2, so this analysis is the same as previously reported; See Primary Objectives for additional details

4. Secondary Outcome: Change in Time to Diagnosis of SND Before and After Intervention
Description: Time to diagnosis days (date of diagnosis - date of enrollment)
Time Frame: From date of enrollment until date of SND diagnosis, assessed up to 60 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 368 | 409
Participants
  0 Months (or Prior to Enrollment) | 126 | 232
  Prior to 1 Month | 168 | 156
  1-2 Months | 10 | 7
  2-3 Months | 7 | 4
  3-4 Months | 6 | 1
  4-5 Months | 2 | 3
  5-6 Months | 2 | 2
  Greater than 6 Months | 47 | 4

5. Secondary Outcome: Change in Time to Receiving an Indicated IPG Device for Subjects Diagnosed With SND Before and After Intervention
Description: Time to implant in days (date of implant - date of diagnosis)
Time Frame: From date of SND diagnosis until date of therapy, assessed up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 | Phase 2
Number analyzed (Participants) | 63 | 130
Participants
  0 Months or Prior to Implant | 22 | 52
  Prior to 1 Month | 37 | 74
  1-2 Months | 1 | 0
  2-3 Months | 0 | 2
  Greater than 3 Months | 3 | 2

6. Secondary Outcome: Difference in QoL Between Implant Visit and 6 Months Post-implant
Description: The difference in quality of life was assessed using the SF-12 survey, with higher numbers indicating a better quality of life for the patient. The possible physical score ranges are between 24.0 and 56.6. The possible mental score ranges are between 19.1 and 60.8. Only the difference over time was reported.
Time Frame: between implant visit and 6 months post-implant
Population: Only subjects receiving a Medtronic device with both Implant and 6 Month data were included
Measure: Mean (Standard Deviation); unit: difference of score on the SF-12 scale
Groups:
- Phase 2 QoL Cohort: Subjects with QoL scores at implant and 6 Months
Arm/Group | Phase 2 QoL Cohort
Number analyzed (Participants) | 69
difference of score on the SF-12 scale
  SF-12 Physical Component | 11.7 (8.1)
  SF-12 Mental Component | 10.2 (10.6)

7. Secondary Outcome: Change in Zarit Quality of Life (QOL) Between Implant Visit and 6 Months Post-implant
Description: The difference in caregiver burden was assessed using a Zarit survey, with lower numbers indicating a decreased burden or a better outcome for the caregiver. The possible range of scores was between 0 and 88. Only the difference in scores over time were reported.
Time Frame: between implant visit and 6 months post-implant
Population: Only subjects receiving a Medtronic device with both Implant and 6 Month data were included
Measure: Mean (Standard Deviation); unit: change in score on Zarit QoL scale
Arm/Group | Phase 2 QoL Cohort
Number analyzed (Participants) | 69
change in score on Zarit QoL scale | -14.7 (15.7)

ADVERSE EVENTS:
Time Frame: Study duration lasted 6 months
Description: Adverse events beyond death were not collected in this study.
Groups:
- Phase I: Characterize the current management of patients presenting with possible sinus node dysfunction
- Phase II: Assess the effect of critical care pathways, education and comprehensive disease state management on the adoption of ACC/AHA/HRS and ESC indications and therapies for sinus node dysfunction.
Arm/Group | Phase I | Phase II
All-Cause Mortality (participants affected / at risk) | 2/847 | 1/470
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Non-randomized observational study, data collected in a limited region with 10 specialized centers.Assumptions on the effect of pacemaker therapy affordability were limited.QoL increases were not compared to an age and gender-matched control group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2012-02-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT01643707/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT01643707/SAP_001.pdf